CLINICAL TRIAL: NCT03667222
Title: PRISM: A Double Blind, Randomized, Vehicle Controlled Phase 2 Study to Assess the Safety and Efficacy of BPX-04 Minocycline Topical Gel in the Treatment of Inflammatory Lesions of Papulopustular Rosacea
Brief Title: Topical Minocycline Gel for Inflammatory Lesions of Papulopustular Rosacea
Acronym: PRISM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BioPharmX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BPX-04-C07
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Papulopustular Rosacea
MeSH Terms: conditions — Rosacea | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Vehicle control is identical to the active product in appearance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BPX-04 Active (Experimental): BPX-04 1% minocycline topical gel
  Interventions: Drug: minocycline topical gel
- BPX-04 Vehicle (Placebo Comparator): BPX-04 topical gel vehicle
  Interventions: Drug: topical gel vehicle

INTERVENTIONS:
Drug: minocycline topical gel — Once daily administration of BPX-04 minocycline gel for 12 weeks
  Arms: BPX-04 Active
Drug: topical gel vehicle — Once daily administration of BPX-04 gel vehicle for 12 weeks
  Arms: BPX-04 Vehicle

SUMMARY:
This is a 12-week, multicenter, double-blind, randomized, two-arm, vehicle controlled study. Subjects will be randomized 1:1 to BPX-04 minocycline topical gel 1% or vehicle. This study will include approximately 176 randomized subjects with inflammatory lesions of papulopustular rosacea on the face, defined by an IGA score of 3 (moderate) or 4 (severe) at Baseline. Subjects will be healthy male or female subjects aged 18 years or older. There will be up to 20 study sites in the USA.

DETAILED DESCRIPTION:
This is a 12-week, multicenter, double-blind, randomized, two-arm, vehicle controlled study. Subjects will be randomized 1:1 to BPX-04 minocycline topical gel 1% or vehicle. This study will include approximately 176 randomized subjects with inflammatory lesions of papulopustular rosacea on the face, defined by an IGA score of 3 (moderate) or 4 (severe) at Baseline. Subjects will be healthy male or female subjects aged 18 years or older. There will be up to 20 study sites in the USA.

Subjects will apply approximately 1 gram of topical gel once each day for a 12 week duration. They will come to the study site at Screening, Baseline, and Weeks 4, 8, and 12 or early termination (ET) for the protocol required efficacy and safety evaluations.

At each visit, efficacy will be assessed by rosacea lesion counts, IGA, PGI-S, PGI-I, CGI-S, CGI-I, RosaQoL, Erythema Assessment Scale, Telangiectasia Assessment Scale and subject satisfaction questionnaire.

Safety will be assessed with vital signs, physical examination, laboratory tests such as clinical hematology and chemistries, investigators' and subjects' assessments of cutaneous tolerability, incidence of minocycline-induced skin hyperpigmentation, incidence of visual disturbances and/or headaches suggestive of pseudotumor cerebri, and incidence of TEAEs. Blood samples will be collected to evaluate the level of minocycline in plasma at Baseline and Week 12/ET.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years of age at the time of consent.
2. Subjects do not have any medical conditions, other than rosacea, that in the opinion of the investigator, put the subject at unacceptable risk or could interfere with study assessments or integrity of the data.
3. A clinical diagnosis of moderate to severe (Grade 3 or 4) facial rosacea (papulopustular (Subtype 2) or mixed erythematotelangiectatic (Subtype 1) and papulopustular (Subtype 2)) as determined by the Investigator's Global Assessment (IGA)
4. Have 15-70 papulopustular lesions of rosacea on the face with no more than 2 nodules.
5. Female subjects of childbearing potential are willing to use effective contraceptive method (s) for at least 4 weeks before Baseline and at least 4 weeks after the last study product administration or have a sterilized or same sex partner for the duration of the study. Effective contraceptive methods are: systemic hormonal contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicide or agree to sexual abstinence. Hormonal contraceptives must be on a stable dose for at least 12 weeks before Baseline. Subjects using low dose (≤35 ug ethinyl estradiol) oral contraceptives must use a second form of birth control (e.g., barrier method such as condoms with spermicide).
6. Female subjects of childbearing potential must have a negative urine pregnancy test (dipstick).
7. Subjects who use make-up, facial moisturizers, creams, lotions, cleansers and/or sunscreens must have used the same product brands/types for a minimum period of 2 weeks prior to Baseline, must agree not to change brand/type or frequency of use throughout the study and must agree not to use make-up, facial moisturizers, creams, lotions, cleansers and/or sunscreens on the scheduled clinic visit days before the visit.
8. Be willing to limit or avoid known personal 'triggers' of rosacea such as spicy foods, consumption of alcoholic beverages, extended sun exposure, tanning beds, etc., for the duration of the study.
9. Subjects must be capable of giving informed consent and the written informed consent must be obtained prior to any study-related procedures.

Exclusion Criteria:

1. Have a history of skin disease, presence of skin condition, scarring or excessive facial hair the PI believes would interfere with the study.
2. Have moderate or severe rhinophyma, severe telangiectasia or plaque-like facial edema.
3. Have rosacea conglobata or fulminans, corticosteroid induced rosacea or facial erythrosis other than rosacea.
4. Have ocular rosacea of a severity that requires systemic treatment.
5. Have a history of any adverse reaction to minocycline or other tetracycline class antibiotic.
6. Have a clinically significant chemistry or hematology value or have an ALT or AST that is greater than or equal to 2x normal.
7. Have any conditions or factors that the PI believes may affect the response of the skin or the interpretation of the results.
8. Have a history of symptoms that might be confused with a diagnosis of pseudotumor cerebri such as severe headaches or visual disturbances inconsistent with a diagnosis of migraine or have a history of traumatic brain injury with headache and/or visual disturbances.
9. Have used on the face an over the counter (OTC) topical medication for the treatment of rosacea within 4 weeks prior to Baseline.
10. Have used prescription topical (on the face) and/or oral antibiotics within 4 weeks prior to Baseline.
11. Treatment with hormonal therapy or oral corticosteroids that is not on a stable dose and frequency for at least 12 weeks before Baseline and not stable throughout the study.
12. Have had a facial procedure such as chemical peel, laser, microdermabrasion or injections with a dermal filler or neuromodulator within 8 weeks prior to Baseline.
13. Have received photodynamic therapy or phototherapy to the face within 12 weeks prior to Baseline.
14. Have used an oral retinoid within 6 months or a topical retinoid within 3 months prior to Baseline.
15. Current drug or alcohol abuse.
16. Female subject who is breastfeeding, pregnant or who is planning a pregnancy during the study.
17. Participated in any clinical study with exposure to any investigational treatment or product within the previous 4 weeks to Baseline, or plan on concurrent participation in other studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-08-17 (Estimated)

PRIMARY OUTCOMES:
Inflammatory lesion count | Baseline to Week 12
  Change in mean facial inflammatory lesion count

SECONDARY OUTCOMES:
Change in IGA | Baseline to Week 12
  Proportion of subjects with ≥2-point change in IGA of rosacea to clear or almost clear

CONTACTS AND LOCATIONS:
Overall Officials: AnnaMarie Daniels, Study Director — BioPharmX, Inc.
Locations (12):
- United States (12):
  - Study Center, Anaheim Hills, California
  - Study Center, Miami, Florida
  - Study Center, Miramar, Florida
  - Study Center, Baton Rouge, Louisiana
  - Study Center, New Orleans, Louisiana
  - Study Center, Needham, Massachusetts
  - Study Center, Saint Joseph, Missouri
  - Study Center, Morristown, New Jersey
  - Study Center, High Point, North Carolina
  - Study Center, Philadelphia, Pennsylvania
  - Study Center, Austin, Texas
  - Study Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No